CLINICAL TRIAL: NCT02398318
Title: China Refractory-Obsessive Compulsive Disorder Deep Brain Stimulation Study
Brief Title: China Refractory Obsessive-Compulsive Disorder Deep Brain Stimulation Study
Acronym: CRODS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: A pilot study is recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Suzhou Sceneray Medical Co. , Ltd (Industry); National Natural Science Foundation of China (Other Government); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of functional neurosurgery department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT-YY2015-CRODS
Record Dates: First submitted 2015-01-23; First posted 2015-03-25 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Obsessive Compulsive Disorder
Keywords: neurosurgery; deep brain stimulation; exposure response prevention
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilateral Nucleus Accumbens DBS (Active Comparator): 6 month period of active bilateral nucleus accumbens DBS
  Interventions: Device: Bilateral Nucleus Accumbens DBS (Suzhou Sceneray)
- Sham Bilateral Nucleus Accumbens DBS (Sham Comparator): 6 month period of sham bilateral nucleus accumbens DBS
  Interventions: Device: Sham Bilateral Nucleus Accumbens DBS

INTERVENTIONS:
Device: Bilateral Nucleus Accumbens DBS (Suzhou Sceneray) — High frequency stimulation applied using Suzhou Sceneray® DBS hardware (1120 electrode, 1180 (S) battery).
  Other Names: Active DBS
  Arms: Bilateral Nucleus Accumbens DBS
Device: Sham Bilateral Nucleus Accumbens DBS — DBS system switched off.
  Other Names: Sham DBS
  Arms: Sham Bilateral Nucleus Accumbens DBS

SUMMARY:
Refractory obsessive-compulsive disorder (OCD) is a disabling condition. Deep brain stimulation (DBS) of the nucleus accumbens is the most tested therapeutic avenue for refractory OCD. However, large scale randomized controlled trials to evaluate the effectiveness of this approach are rare.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. A primary diagnosis of OCD, defined according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV).
3. Chronic: disease duration of more than 5 years.
4. Severity: a score on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) of more than 25 or one subscale score of more than 15 ; a score for severity of illness on the Clinical Global Impression (CGI) scale of more than 4.
5. Disability: a score on the Global Assessment Functioning (GAF) scale of less than 45.
6. Refractory: a lack of response to drug therapy after adequate administration (defined as more than 12 weeks at the maximum tolerated dose) of at least three serotonin-reuptake inhibitors, one of which had to be clomipramine. Adequate behavior therapy, defined as 20 sessions of exposure and response prevention (ERP) with a therapist who has substantial expertise in OCD treatment.

Exclusion Criteria:

1. Schizophrenic disorder; bipolar disorder; substance abuse or dependence (except for dependence on nicotine), as assessed with the use of the Mini-International Neuropsychiatric Interview (MINI 6.0.0).
2. Cluster A or B personality disorder according to DSM-IV criteria, as assessed with the use of the Structured Clinical Interview II.
3. A current severe major depressive episode, determined according to DSM-IV criteria (as assessed with the use of the MINI 6.0.0) and defined by the Hamilton Depression Rating Scale-17 (HAMD) score of more than 20 and a risk of suicide.
4. Abnormal cognitive status (measured by MoCA), abnormal findings on functional magnetic resonance imaging (MRI) of the brain; and no contraindications to surgery or anesthesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) Score | Baseline (preoperative), 6 months

SECONDARY OUTCOMES:
Change in Obsessive-Compulsive Inventory - Revised (OCI-R) Score | Baseline (preoperative), 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months
Change in Hamilton Anxiety Scale, Hamilton Depression Scale-17, Beck Anxiety Scale, Beck Depression Scale-1 Score | Baseline (preoperative), 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months
Change in Temperament and Character Inventory revised version (TCI-R) Score | Baseline (preoperative), 6 months, 24 months
Iowa Gambling Task (change in task performance scores) | Baseline (preoperative), 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months
Change in functional magnetic resonance imaging (fMRI) images | Baseline (preoperative), 2 weeks after last ERP session (average)
Change in positron emission tomography (PET) brain glucose metabolism images | Baseline (preoperative), 6 months after surgery
  Fluoro-D-glucose (FDG) will be utilized to evaluate cerebral metabolism at Baseline (preoperative) and 6 months.
Quality of life: Global assessment of function | Baseline (preoperative), 2 weeks after last ERP session (average), 6 months after surgery, 24 months after surgery
Disability: WHO disability assessment 2.0 | Baseline (preoperative), 2 weeks after last ERP session (average), 6 months after surgery, 24 months after surgery
Model Task (change in task performance scores) | Baseline (preoperative), 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, MD,PhD, Principal Investigator — Ruijin Hospital
Locations (3):
- China (3):
  - Guangzhou psychiatric hospital, Guangzhou, Guangdong
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan

REFERENCES:
- [Background] Zuo C, Ma Y, Sun B, Peng S, Zhang H, Eidelberg D, Guan Y. Metabolic imaging of bilateral anterior capsulotomy in refractory obsessive compulsive disorder: an FDG PET study. J Cereb Blood Flow Metab. 2013 Jun;33(6):880-7. doi: 10.1038/jcbfm.2013.23. Epub 2013 Feb 27. PMID 23443174
- [Background] Wu H, Van Dyck-Lippens PJ, Santegoeds R, van Kuyck K, Gabriels L, Lin G, Pan G, Li Y, Li D, Zhan S, Sun B, Nuttin B. Deep-brain stimulation for anorexia nervosa. World Neurosurg. 2013 Sep-Oct;80(3-4):S29.e1-10. doi: 10.1016/j.wneu.2012.06.039. Epub 2012 Jun 25. PMID 22743198
- [Derived] Xiong B, Li B, Wen R, Gao Y, Gong F, Li D, Xu Y, Deng H, Xiao L, Yin S, Zhang W, Lozano AM, Wang W. Use of differential stimulation of the nucleus accumbens and anterior limb of the internal capsule to improve outcomes of obsessive-compulsive disorder. J Neurosurg. 2023 May 26;139(5):1376-1385. doi: 10.3171/2023.4.JNS221824. Print 2023 Nov 1. PMID 37243560
- See also: Related Info — http://www.mitoonet.com/rjh